CLINICAL TRIAL: NCT00373633
Title: A Prospective Randomized Trial Comparing Extrapleural Intercostal Local Anesthesia Versus Thoracic Epidural for the Managment of Acute Post Thoracotomy Pain
Brief Title: Extrapleural Intercostal Catheter vs. Thoracic Epidural for Thoracotomy Pain
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: terminated due to diminishing frequency of thorocotomies and slow enrollment
Sponsor: Virginia Commonwealth University (Other)
Collaborators: I-Flow (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: VCU 011906
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: THoracotomy
Keywords: THoracic Surgery; thoracic epidural; epidural; thoracotomy; intercostal nerve block; intercostal; nerve block
MeSH Terms: interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Continuous extra-pleural intercostal local anesthesia (Experimental): intra-operatively placed extrapleural intercostal catheter
  Interventions: Procedure: Extrapleural Intercostal Catheter
- Thoracic Epidural (Active Comparator): gold standard
  Interventions: Procedure: Thoracic Epidural

INTERVENTIONS:
Procedure: Thoracic Epidural — Gold standard for post thoracotomy pain
  Arms: Thoracic Epidural
Procedure: Extrapleural Intercostal Catheter — Continuous extra-pleural intercostal local anesthesia
  Arms: Continuous extra-pleural intercostal local anesthesia

SUMMARY:
We will compare thoracic epidural anesthesia which is presently used for management of pain after thoracotomy to an intra-operatively placed extrapleural intercostal catheter. The study wil be double blinded and prospective.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy of thoracic epidural vs. continuous extra-pleural intercostal local anesthesia for the treatment of post thoracotomy pain in adult patients. Study patients will be randomized between the thoracic epidural and continuous extrapleural catheter groups[Figure 1]. Because thoracic epidural anesthesia is the gold standard but continuous extrapleural intercostal local anesthesia is potentially easier and less prone to complications, the study will be structured as an "equivalence study". The null hypothesis (Ho) is that continuous intercostal nerve blockade is worse than epidural for post-thoracotomy pain management. Therefore, the alternative hypothesis (Ha) is then that continuous intercostal nerve blockade is equal to or better than epidural for post-thoracotomy pain management.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral thoracotomy
* Video Assisted thoracotomy with high likely hood of converting to open thoracotmoy

Exclusion Criteria:

* Bilateral thoracotomy
* Planned bilateral thoracotomy
* Planned chest wall resection
* Planned combined thoracotomy and laparotomy procedure
* VATS procedure without conversion to unilateral thoracotomy
* Emergency operation
* Critically ill patients
* Patients who require an assistive device (i.e. cane, walker, or wheel chair) for mobility
* Patients who are unable to give informed consent
* Patients with preoperative chronic back or chest wall pain
* Empyema or other infective condition increasing the risk of epidural infection
* Coagulopathy
* Decision of the surgeon or anesthesiologist, or choice of the patient
* Infection at site of epidural placement
* Patients with other co morbidities which exclude thoracic epidural placement
* Patients under the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
pain control-visual analog pain score | post surgery monitoring

SECONDARY OUTCOMES:
respiratory measurements (FEV1, PEF), pain score, nausea and vomiting, opiod usage as adjunct to primary treatmetn modalities | post surgery monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nelson, MD, Principal Investigator — Virgina Commonwealth University, Dept of Anesthesia
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States